CLINICAL TRIAL: NCT00864123
Title: D-Cycloserine Augmentation of Therapy for Pediatric Obsessive-Compulsive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Principal Investigator, Eric Storch, Associate Professor, University of South Florida
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MH076775; MH076775
Record Dates: First submitted 2009-03-17; First posted 2009-03-18 (Estimated); Results first posted 2012-10-17 (Estimated); Last update posted 2012-10-17 (Estimated); Status verified 2012-09

CONDITIONS: Obsessive-compulsive Disorder
Keywords: Obsessive-compulsive disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Cognitive Behavioral Therapy; Cycloserine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive-behavioral therapy + placebo (Active Comparator): Involves receiving cognitive-behavioral treatment of OCD symptoms for 10 sessions. One hour prior to sessions 4-10, the child will take either 1 or 2 pills containing 25mg of placebo. The number of pills depends on the child's weight (e.g., about 46kgs takes 2 capsules).
  Interventions: Behavioral: Cognitive-behavioral therapy; Drug: Placebo pill
- Cognitive-behavioral therapy + D-cycloserine (Experimental): Involves receiving cognitive-behavioral treatment of OCD symptoms for 10 sessions. One hour prior to sessions 4-10, the child will take either 1 or 2 pills containing 25mg of D-cycloserine. The number of pills depends on the child's weight (e.g., about 46kgs takes 2 capsules).
  Interventions: Behavioral: Cognitive-behavioral therapy; Drug: D-cycloserine

INTERVENTIONS:
Behavioral: Cognitive-behavioral therapy — All patients will receive 10 sessions of therapy over 8 weeks that is based on the protocol used in POTS (2004). Sessions 1-4 will be held twice weekly; thereafter sessions will be held on a weekly basis. This evidence-based E/RP intervention (POTS, 2004) includes psychoeducation, cognitive training, and exposure and response prevention. By design, this manual provides sufficient flexibility to accommodate the child's developmental needs and address maladaptive parent-child interactions (e.g., accommodation).
Drug: D-cycloserine — D-cycloserine (Seromycin, 250 mg; Eli Lilly and Co, Indianapolis, Indiana) will be capsulated into 25mg with identical placebo capsules. Children weighing between 25-45kg will be given a dosage of 25mg (approximately 0.56-1.0 mg/kg/day). Children weighing between 46-80kg will be given a dosage of 50mg (approximately 0.63-1.08mg/kg/day). DCS or placebo will be given by parents 1 hour prior to psychotherapy sessions (before sessions 4-10 only) based on past success in patients with acrophobia (Ressler et al., 2004) and DCS absorption rates.
  Other Names: Seromycin; d-4-amino-3-isoxazolidone
  Arms: Cognitive-behavioral therapy + D-cycloserine
Drug: Placebo pill — This intervention involves taking a placebo pill(s) that matches the d-cycloserine capsules in size, shape, weight, and taste. Placebo contains an no active medication.
  Other Names: Pill placebo
  Arms: Cognitive-behavioral therapy + placebo

SUMMARY:
Cognitive-behavioral therapy (CBT) has proven efficacy for treatment of pediatric obsessive-compulsive disorder (OCD). Yet, CBT does not help all children and those who benefit often remain symptomatic upon treatment completion. Recent clinical trials in adults with other anxiety disorders (acrophobia and social phobia) provided support for using a medication called D-Cycloserine (DCS) to enahnce the outcome of exposure-based psychotherapy. Given this, DCS may augment CBT in youth with OCD, an anxiety disorder that is conceptually similar to acrophobia. With this in mind, the investigators are conducting a randomized, double-blind placebo controlled pilot study of DCS to determine whether it had any short-term clinical benefits on CBT in youth with OCD. Forty children and adolescents (ages 8-17) with a primary diagnosis of OCD will be screened and, should they meet relevant criteria, randomly assigned to one of two treatment conditions: (1) CBT plus DCS, or (2) CBT plus placebo. All patients will receive 10 sessions of CBT A rater will assess participants at 3 separate time points.

DETAILED DESCRIPTION:
Cognitive-behavioral therapy (CBT) has proven efficacy for treatment of pediatric obsessive-compulsive disorder (OCD). Yet, CBT does not help all children and those who benefit often remain symptomatic upon treatment completion. The behavioral theory that underlies CBT is based on two components, namely fear conditioning and extinction. On a neural level, CBT incorporates similar mechanisms to those involved in fear conditioning. Antagonists at the N-methyl-D-aspartate (NMDA) glutamatergic receptor, which is involved in learning and memory, block both fear learning and extinction. Evidence suggests that D-Cycloserine (DCS), a partial agonist at the NMDA glutamate receptor, augments associative learning and extinction as a form of learning in animals and humans. Recent clinical trials in adults with other anxiety disorders (acrophobia and social phobia) provided support for DCS dosing as facilitating associative learning that occurs during exposure-based psychotherapy. Given that CBT is based on the principles of extinction, DCS may augment CBT in youth with OCD, an anxiety disorder that is conceptually similar to acrophobia. With this in mind, I propose to undertake a randomized, double-blind placebo controlled pilot study of DCS to determine whether it had any short-term clinical benefits on CBT in youth with OCD. Forty children and adolescents (ages 8-17) with a primary diagnosis of OCD will be screened and, should they meet relevant criteria, randomly assigned to one of two treatment conditions: (1) CBT plus DCS (25 or 50mg depending on weight), or (2) CBT plus placebo. All patients will receive 10 sessions of CBT based on the protocol used in POTS (2004). Participants will take DCS or placebo 1 hour prior to each therapy session. A blinded, independent evaluator will assess participants at 3 separate time points. Two of the assessments (Baseline, Post-treatment) will be comprehensive in nature (e.g., diagnostic interview, self-reports, CY-BOCS, laboratory tests), whereas one midpoint assessment will involve administration of CY-BOCS, CGI, CGI-S, and Adverse Symptom Checklist only. Results from this study may have powerful clinical implications by providing preliminary support for pharmalogical agents that enhance the effectiveness of standard E/RP. Such agents may have utility in improving outcome, reducing premature therapy termination, and targeting patients who have been treatment refractory.

ELIGIBILITY:
Inclusion Criteria:

* The child must receive a principal diagnosis of OCD at Baseline, based on DSM-IV criteria. This diagnosis will be derived from the Anxiety Disorder Interview Schedule for DSM-IV-Child Interview Schedule - Parent version (ADIS-IV-P), and must reflect a clinical severity rating of 4 or above
* CY-BOCS Total Score ≥ 16
* Be between the ages of 8 and 17 years
* Score ≥ 80 on the Peabody Picture Vocabulary Test-3rd Edition (Dunn & Dunn, 1997)
* At least one parent available to accompany the child to all sessions;
* English speaking.

Exclusion Criteria:

* Psychosis, pervasive developmental disorder, bipolar disorder, or current suicidal intent measured by the ADIS-IV-P and all available clinical information
* Principal diagnosis other than OCD
* Youth with mental rituals, incompleteness, or hoarding symptoms as E/RP exercises would be more difficult to conduct/monitor than those with overt rituals
* Unavailability of at least one caregiver to participate in the treatment
* Refusal of parent to accept random assignment to treatment condition
* A positive diagnosis in the caregiver of mental retardation, psychosis, clinically significant tics, or other psychiatric disorders or conditions that would limit their ability to understand E/RP (based on clinical interview)
* Weight less than 25.0 kg or greater than 80.0kg
* Epilepsy, renal insufficiency, and current or past history of alcohol abuse (DCS is contraindicated for such conditions)
* Pregnant or having unprotected sex [in females] as the effects of DCS on pregnant youth are unknown
* General poor physical health as determined by medical physical and laboratory tests.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2008-01; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Storch, Ph.D., Principal Investigator — University of South Florida
Locations (1):
- University of South Florida, St. Petersburg, Florida, United States

REFERENCES:
- [Result] Storch EA, Murphy TK, Goodman WK, Geffken GR, Lewin AB, Henin A, Micco JA, Sprich S, Wilhelm S, Bengtson M, Geller DA. A preliminary study of D-cycloserine augmentation of cognitive-behavioral therapy in pediatric obsessive-compulsive disorder. Biol Psychiatry. 2010 Dec 1;68(11):1073-6. doi: 10.1016/j.biopsych.2010.07.015. PMID 20817153
- [Derived] Guzick AG, Geller DA, Small BJ, Murphy TK, Wilhelm S, Storch EA. Irritability in Children and Adolescents With OCD. Behav Ther. 2021 Jul;52(4):883-896. doi: 10.1016/j.beth.2020.11.001. Epub 2020 Nov 12. PMID 34134828
- [Derived] Storch EA, McGuire JF, Schneider SC, Small BJ, Murphy TK, Wilhelm S, Geller DA. Sudden gains in cognitive behavioral therapy among children and adolescents with obsessive compulsive disorder. J Behav Ther Exp Psychiatry. 2019 Sep;64:92-98. doi: 10.1016/j.jbtep.2019.03.003. Epub 2019 Mar 9. PMID 30877851
- [Derived] Wilhelm S, Berman N, Small BJ, Porth R, Storch EA, Geller D. D-Cycloserine augmentation of cognitive behavior therapy for pediatric OCD: Predictors and moderators of outcome. J Affect Disord. 2018 Dec 1;241:454-460. doi: 10.1016/j.jad.2018.07.042. Epub 2018 Jul 20. PMID 30149332
- [Derived] Storch EA, Wilhelm S, Sprich S, Henin A, Micco J, Small BJ, McGuire J, Mutch PJ, Lewin AB, Murphy TK, Geller DA. Efficacy of Augmentation of Cognitive Behavior Therapy With Weight-Adjusted d-Cycloserine vs Placebo in Pediatric Obsessive-Compulsive Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2016 Aug 1;73(8):779-88. doi: 10.1001/jamapsychiatry.2016.1128. PMID 27367832

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Excluded (n = 22) Not interested in participating in study (n=9) Changing medication at Baseline (n=5) Did not receive at least one DCS dose (n = 4) History of adequate CBT course (n=2) Met criteria for comorbid autism (n=1) Did not show up for pre-treatment assessment (n=1)
Period: Overall Study
Arm/Group | Cognitive-behavioral Therapy + Placebo | Cognitive-behavioral Therapy + D-cycloserine
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive-behavioral Therapy + Placebo | Cognitive-behavioral Therapy + D-cycloserine | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15 | 15 | 30
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 12.5 (3.5) | 11.9 (1.9) | 12.2 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 9 | 10 | 19
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Children's Yale-Brown Obsessive-Compulsive Scale (CY-BOCS; Scahill et al., 1997).
Description: The CY-BOCS is a 10-item semi-structured measure of obsession and compulsion severity over the previous week. This measure served as the primary outcome index. Scores range from 0-40 with higher scores representing more severe symptoms.
Time Frame: Baseline, Mid-Treatment, Post-treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive-behavioral Therapy + Placebo | Cognitive-behavioral Therapy + D-cycloserine
Number analyzed (Participants) | 15 | 15
units on a scale
  Baseline | 26 (3.8) | 24.1 (4.4)
  Mid-treatment | 17.9 (4.5) | 15.6 (6.8)
  Post-treatment | 11 (6.6) | 6.8 (6)
Statistical Analysis 1: Comparison: Cognitive-behavioral Therapy + Placebo vs Cognitive-behavioral Therapy + D-cycloserine; Data were analyzed with separate 2 (site: Florida, MGH) by 2 (condition: CBT+DCS, CBT+Placebo) by 3 (time: pre-treatment, mid-treatment, post-treatment; Dependent variables: CY-BOCS Total Score) fixed-effects linear regression with time as the repeated measure. Cohen's d was used to examine the magnitude of treatment effects; Test type: Superiority or Other; p < 0.05, ANOVA; Mean Difference (Final Values) = 11.0, Standard Deviation 6.3

2. Secondary Outcome: Clinical Global Impression - Severity (CGI-S; National Institute of Mental Health, 1985). The CGI-S is a 7-point Clinician Rating of Severity of Psychopathology.
Description: The CGI-S is a 7-point clinician rating of severity of psychopathology. Ratings range from 1 ("no illness") to 7 ("extremely severe"). A single rating is chosen for the CGI-S; thus, there are no summary scales/scores.
Time Frame: Baseline, mid-treatment, post-treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive-behavioral Therapy + Placebo | Cognitive-behavioral Therapy + D-cycloserine
Number analyzed (Participants) | 15 | 15
units on a scale
  Baseline | 5.1 (.74) | 4.6 (.83)
  Mid-treatment | 3.9 (.59) | 3.5 (.92)
  Post-treatment | 3 (1.2) | 2 (1)
Statistical Analysis 1: Comparison: Cognitive-behavioral Therapy + Placebo vs Cognitive-behavioral Therapy + D-cycloserine; Data were analyzed with separate 2 (site: Florida, MGH) by 2 (condition: CBT+DCS, CBT+Placebo) by 3 (time: pre-treatment, mid-treatment, post-treatment; Dependent variables: CGI-Severity) fixed-effects linear regression with time as the repeated measure. Cohen's d was used to examine the magnitude of treatment effects; Test type: Superiority or Other; p < 0.05, ANOVA; Mean Difference (Final Values) = 3, Standard Deviation 1.1

3. Secondary Outcome: Adverse Symptom Checklist (ASC; Goodman, 2005).
Description: This index assesses adverse side effects that have been associated with DCS, as well as other commonly used psychotropic agents (e.g., SRIs). There are no summary scales for this. Rather, it reflects the presence or absence of 30 potential side effects on a 0-3 scale (0=not at all, 1=slight, 2=moderate, 3=severe) that are associated with study interventions.
Time Frame: Baseline, mid-treatment, post-treatment
Population: Number of participants experiencing an adverse effect related to study interventions. This is a simple frequency count.
Measure: Number; unit: participants
Arm/Group | Cognitive-behavioral Therapy + Placebo | Cognitive-behavioral Therapy + D-cycloserine
Number analyzed (Participants) | 15 | 15
participants
  Baseline | 0 | 0
  Mid-treatment | 0 | 0
  Post-treatment | 0 | 0

ADVERSE EVENTS:
Description: This metric refers to the number of youth experiencing an adverse event associated with study interventions.
Arm/Group | Cognitive-behavioral Therapy + Placebo | Cognitive-behavioral Therapy + D-cycloserine
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No